CLINICAL TRIAL: NCT07352839
Title: Comparison of Brachial Plexus Block Versus General Anesthesia for Upper Extremity Surgery: A Randomized Controlled Trial
Brief Title: Brachial Plexus Block vs General Anesthesia in Upper Extremity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek Uçak, Principal Investigator, Department of Anesthesiology and Reanimation, Adana City Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 536
Record Dates: First submitted 2025-12-30; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Upper Extremity Surgery; Regional Anesthesia; General Anesthetic
MeSH Terms: interventions — Brachial Plexus Block; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brachial Plexus Block Group (Active Comparator): Patients receiving ultrasound-guided brachial plexus block for upper extremity surgery
  Interventions: Procedure: Brachial Plexus Block
- General Anesthesia Group (Active Comparator): Patients receiving general anesthesia for upper extremity surgery
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Brachial Plexus Block — Ultrasound-guided infraclavicular brachial plexus block using local anesthetic (e.g., ropivacaine or bupivacaine). Block performed before surgery to provide regional anesthesia for upper extremity surgery.
  Arms: Brachial Plexus Block Group
Procedure: General Anesthesia — Standard general anesthesia with intravenous induction and maintenance with volatile anesthetics or total intravenous anesthesia (TIVA). Endotracheal intubation or laryngeal mask airway used as appropriate.
  Arms: General Anesthesia Group

SUMMARY:
This study compares two different anesthesia methods for upper arm and hand surgery: regional anesthesia (brachial plexus block) versus general anesthesia.

Regional anesthesia numbs only the arm being operated on by injecting local anesthetic near the nerves, while the patient remains awake or lightly sedated. General anesthesia puts the patient completely asleep using medications given through a breathing tube.

The main goals of this study are to compare:

* How much pain patients experience after surgery
* Patient satisfaction with their anesthesia
* Side effects such as nausea, vomiting, or breathing problems
* Time until patients are ready to go home
* Overall safety of each method

Participants in this study will be randomly assigned to receive either brachial plexus block or general anesthesia for their scheduled upper extremity surgery. The research team will monitor participants during surgery and follow their recovery for 24 hours after the operation.

This research will help doctors and patients make better-informed decisions about which type of anesthesia may be best for upper extremity procedures.

ELIGIBILITY:
Inclusion Criteria:

* clusion Criteria:
* Adults aged 18-65 years
* ASA physical status I-II
* Scheduled for elective upper-extremity orthopedic surgery
* Able to provide informed consent
* Able to understand and complete study questionnaires

Exclusion Criteria:

* Contraindications to regional anesthesia
* Coagulopathy or bleeding disorders
* Local infection at the block site
* Patient refusal of regional anesthesia
* Known allergy to local anesthetic agents
* Chronic opioid use (daily use for >3 months)
* Psychiatric disorders preventing cooperation or consent
* Pregnancy or breastfeeding
* Severe respiratory disease (for general anesthesia group)
* Pre-existing neurological deficit in the operative extremity
* Emergency surgery
* ASA physical status III or higher

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Preoperative Anxiety Score | Immediately before operating room entry (preoperatively)
  Preoperative anxiety measured immediately prior to operating room entry using the State-Trait Anxiety Inventory-State (STAI-S) scale. STAI-S is a validated 20-item questionnaire assessing current state anxiety. Scores range from 20 to 80, with higher scores indicating greater anxiety levels.

SECONDARY OUTCOMES:
Postoperative Pain Score | From end of surgery to 24 hours postoperatively
  Pain intensity measured using Visual Analog Scale (VAS) at multiple time points after surgery. VAS scores range from 0 to 10, where 0 indicates no pain and 10 indicates worst pain imaginable. Lower scores indicate better outcome.
Opioid Consumption | From end of surgery to 24 hours postoperatively
  Total opioid consumption measured as morphine equivalent dose (mg) during the postoperative period. All opioid medications administered were converted to morphine equivalents using standard conversion factors. Lower consumption indicates better outcome.
Number of Participants with Postoperative Nausea and Vomiting (PONV) | First 24 hours postoperatively
  Number of participants experiencing postoperative nausea and/or vomiting requiring antiemetic treatment during the postoperative period. PONV was defined as any episode of nausea or vomiting reported by the patient or requiring rescue antiemetic medication.
PACU Length of Stay | From PACU admission until discharge readiness (typically 0-4 hours postoperatively
  Duration of stay in the Post-Anesthesia Care Unit (PACU) measured in minutes, from admission to discharge readiness based on standardized discharge criteria (Aldrete score ≥9). Shorter stay indicates better recovery.
Quality of Recovery (QoR-15) Score | 24 hours postoperatively
  Patient-reported quality of recovery assessed using the validated Quality of Recovery-15 (QoR-15) questionnaire. QoR-15 is a 15-item instrument measuring five dimensions of recovery: physical comfort, emotional state, psychological support, physical independence, and pain. Each item is scored 0-10, with total scores ranging from 0 to 150. Higher scores indicate better quality of recovery.
Patient Satisfaction Score | 24 hours postoperatively
  Overall patient satisfaction with anesthesia care measured using a numerical rating scale from 0 to 5, where 0 indicates completely dissatisfied and 5 indicates completely satisfied. Patients were asked to rate their overall satisfaction with the anesthesia experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Adana City Training and Research Hospital, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No